CLINICAL TRIAL: NCT02477826
Title: An Open-Label, Randomized Phase 3 Trial of Nivolumab, or Nivolumab Plus Ipilimumab, or Nivolumab Plus Platinum Doublet Chemotherapy Versus Platinum Doublet Chemotherapy in Subjects With Chemotherapy-Naïve Stage IV or Recurrent Non-Small Cell Lung Cancer (NSCLC)
Brief Title: An Investigational Immuno-therapy Trial of Nivolumab, or Nivolumab Plus Ipilimumab, or Nivolumab Plus Platinum-doublet Chemotherapy, Compared to Platinum Doublet Chemotherapy in Patients With Stage IV Non-Small Cell Lung Cancer (NSCLC)
Acronym: CheckMate 227
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: Ono Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA209-227; 2014-003630-23 (EudraCT Number)
Record Dates: First submitted 2015-06-18; First posted 2015-06-23 (Estimated); Results first posted 2025-10-30 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Nivolumab; Ipilimumab; Carboplatin; Cisplatin; Gemcitabine; Pemetrexed; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Arm A: Nivolumab (Experimental): Nivolumab intravenously (IV) as specified
  Interventions: Drug: Nivolumab
- Arm B: Nivolumab + Ipilimumab (Experimental): Nivolumab + Ipilimumab IV as specified
  Interventions: Drug: Nivolumab; Drug: Ipilimumab
- Arm C: Nivolumab + Platinum doublet chemotherapy (Experimental): Nivolumab + Platinum doublet chemotherapy (IV) dose as specified
  Interventions: Drug: Nivolumab; Drug: Carboplatin; Drug: Cisplatin; Drug: Gemcitabine; Drug: Pemetrexed; Drug: Paclitaxel
- Arm D: Platinum doublet chemotherapy (Experimental): Chemotherapy administered on specified days of IV chemotherapy
  Interventions: Drug: Carboplatin; Drug: Cisplatin; Drug: Gemcitabine; Drug: Pemetrexed; Drug: Paclitaxel

INTERVENTIONS:
Drug: Nivolumab
  Other Names: Opdivo
  Arms: Arm A: Nivolumab; Arm B: Nivolumab + Ipilimumab; Arm C: Nivolumab + Platinum doublet chemotherapy
Drug: Ipilimumab
  Other Names: Yervoy
  Arms: Arm B: Nivolumab + Ipilimumab
Drug: Carboplatin
  Arms: Arm C: Nivolumab + Platinum doublet chemotherapy; Arm D: Platinum doublet chemotherapy
Drug: Cisplatin
  Arms: Arm C: Nivolumab + Platinum doublet chemotherapy; Arm D: Platinum doublet chemotherapy
Drug: Gemcitabine
  Arms: Arm C: Nivolumab + Platinum doublet chemotherapy; Arm D: Platinum doublet chemotherapy
Drug: Pemetrexed
  Arms: Arm C: Nivolumab + Platinum doublet chemotherapy; Arm D: Platinum doublet chemotherapy
Drug: Paclitaxel
  Arms: Arm C: Nivolumab + Platinum doublet chemotherapy; Arm D: Platinum doublet chemotherapy

SUMMARY:
The purpose of this study is to show that Nivolumab, or Nivolumab plus Ipilimumab, or Nivolumab plus Platinum-Doublet Chemotherapy improves progression free survival and/or overall survival compared with chemotherapy in patients with advanced lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with histologically confirmed Stage IV or recurrent NSCLC squamous or non-squamous histology, with no prior systemic anticancer therapy
* Subjects must have programmed death-ligand 1 (PD -L1) immunohistochemical (IHC) testing, with results, performed by the central lab during the Screening period
* Eastern Cooperative Oncology Group (ECOG) Performance Status of ≤ 1
* Measurable disease by CT or MRI per response evaluation criteria in solid tumors version 1.1 (RECIST 1.1) criteria

Exclusion Criteria:

* Subjects with untreated Central nervous system (CNS) metastases are excluded
* Subjects with an active, known or suspected autoimmune disease are excluded
* Any positive test for hepatitis B virus or hepatitis C virus or human immunodeficiency virus (HIV) indicating acute or chronic infection

Other protocol defined inclusion/exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2747 (Actual)
Dates: Start 2015-08-05 (Actual); Primary Completion 2024-10-25 (Actual); Study Completion 2024-10-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (290):
- United States (25):
  - Southern Cancer Center, Inc., Mobile, Alabama
  - Local Institution - 0017, San Francisco, California
  - Local Institution - 0021, New Haven, Connecticut
  - Local Institution - 0001, Atlanta, Georgia
  - Local Institution - 0013, Marietta, Georgia
  - Local Institution - 0004, Lexington, Kentucky
  - Local Institution - 0115, St Louis, Missouri
  - Local Institution - 0005, Buffalo, New York
  - Local Institution - 0019, New York, New York
  - Local Institution - 0014, Cleveland, Ohio
  - Local Institution - 0009, Columbus, Ohio
  - Local Institution - 0007, Allentown, Pennsylvania
  - Local Institution - 0075, Langhorne, Pennsylvania
  - Local Institution - 0299, Philadelphia, Pennsylvania
  - Local Institution - 0012, Philadelphia, Pennsylvania
  - Local Institution - 0015, Sayre, Pennsylvania
  - Local Institution - 0008, Charleston, South Carolina
  - Local Institution - 0080, Greenville, South Carolina
  - Local Institution - 0010, Greenville, South Carolina
  - Local Institution - 0020, Nashville, Tennessee
  - Local Institution - 0306, Dallas, Texas
  - Local Institution - 0003, Dallas, Texas
  - Local Institution - 0102, Houston, Texas
  - Local Institution - 0011, Salt Lake City, Utah
  - Local Institution - 0074, Kennewick, Washington
- Argentina (10):
  - Local Institution - 0170, Berazategui, Buenos Aires
  - Local Institution - 0171, Capital Federal, Buenos Aires
  - Local Institution - 0172, Ciudad Autonoma de Buenos Aire, Buenos Aires
  - Local Institution - 0176, Ciudad de Buenos Aires, Buenos Aires
  - Local Institution - 0296, Mar del Plata, Buenos Aires
  - Local Institution - 0130, San Miguel de Tucumán, Tucumán Province
  - Local Institution - 0268, Córdoba
  - Local Institution - 0272, Córdoba
  - Local Institution - 0297, Córdoba
  - Local Institution - 0177, Viedma
- Australia (10):
  - Local Institution - 0182, Garran, Australian Capital Territory
  - Local Institution - 0301, Blacktown, New South Wales
  - Local Institution - 0300, Gosford, New South Wales
  - Local Institution - 0045, Brisbane, Queensland
  - Local Institution - 0046, Elizabeth Vale, South Australia
  - Local Institution - 0043, Clayton, Victoria
  - Local Institution - 0042, Fitzroy, Victoria
  - Local Institution - 0180, Perth, Western Australia
  - Local Institution - 0040, Murdoch
  - Local Institution - 0183, North Tamworth
- Austria (3):
  - Local Institution - 0241, Graz
  - Local Institution - 0240, Vienna
  - Local Institution - 0239, Wels
- Belgium (6):
  - Local Institution - 0034, Charleroi, Hainaut
  - Local Institution - 0121, Roeselare, West-Vlaanderen
  - Local Institution - 0030, Edegem
  - Local Institution - 0031, Ghent
  - Local Institution - 0117, Hasselt
  - Local Institution - 0033, Sint-Niklaas
- Brazil (8):
  - Local Institution - 0125, Salvador, Estado de Bahia
  - Local Institution - 0124, Ijuí, Rio Grande do Sul
  - Local Institution - 0123, Porto Alegre, Rio Grande do Sul
  - Local Institution - 0127, Barretos, São Paulo
  - Local Institution - 0129, Rio de Janeiro
  - Local Institution - 0144, São Paulo
  - Local Institution - 0126, São Paulo
  - Local Institution - 0128, São Paulo
- Canada (9):
  - Local Institution - 0103, Edmonton, Alberta
  - Local Institution - 0290, St. John's, Newfoundland and Labrador
  - Local Institution - 0104, London, Ontario
  - Local Institution - 0122, Montreal, Quebec
  - Local Institution - 0106, Québec, Quebec
  - Local Institution - 0302, Québec, Quebec
  - Local Institution - 0107, Rimouski, Quebec
  - Local Institution - 0291, Sherbrooke, Quebec
  - Local Institution - 0292, Trois-Rivières, Quebec
- Chile (3):
  - Local Institution - 0174, Viña del Mar, Región de Valparaíso
  - Local Institution - 0173, Santiago, Santiago Metropolitan
  - Local Institution - 0131, Santiago, Santiago Metropolitan
- China (37):
  - Local Institution - 0380, Hefei, Anhui
  - Local Institution - 0313, Beijing, Beijing Municipality
  - Local Institution - 0315, Beijing, Beijing Municipality
  - Local Institution - 0316, Beijing, Beijing Municipality
  - Local Institution - 0314, Beijing, Beijing Municipality
  - Local Institution - 0365, Chongqing, Chongqing Municipality
  - Local Institution - 0364, Chongqing, Chongqing Municipality
  - Local Institution - 0378, Chongqing, Chongqing Municipality
  - Local Institution - 0322, Guangzhou, Guangdong
  - Local Institution - 0372, Guangzhou, Guangdong
  - Local Institution - 0319, Guanzhou, Guangdong
  - Local Institution - 0323, Haikou, Hainan
  - Local Institution - 0325, Haerbin, Heilongjiang
  - Local Institution - 0324, Zhengzhou, Henan
  - Local Institution - 0379, Zhengzhou, Henan
  - Local Institution - 0375, Wuhan, Hubei
  - Local Institution - 0362, Changsha, Hunan
  - Local Institution - 0347, Nanchang, Jiangxi
  - Local Institution - 0329, Changchun, Jilin
  - Local Institution - 0361, Changchun, Jilin
  - Local Institution - 0359, Shenyang, Liaoning
  - Local Institution - 0371, Xi'an, Shaanxi
  - Local Institution - 0333, Xi'an, Shan3xi
  - Local Institution - 0360, Qingdao, Shandong
  - Local Institution - 0336, Shanghai, Shanghai Municipality
  - Local Institution - 0334, Shanghai, Shanghai Municipality
  - Local Institution - 0376, Chengdu, Sichuan
  - Local Institution - 0373, Tianjin, Tianjin Municipality
  - Local Institution - 0340, Ürümqi, Xinjiang
  - Local Institution - 0343, Hangzhou, Zhejiang
  - Local Institution - 0370, Hangzhou, Zhejiang
  - Local Institution - 0342, Hangzhou, Zhejiang
  - Local Institution - 0328, Changsha
  - Local Institution - 0341, Hangzhou
  - Local Institution - 0345, Kunming
  - Local Institution - 0337, Shanghai
  - Local Institution - 0374, Shantou
- Colombia (4):
  - Local Institution - 0273, Pereira, Risaralda Department
  - Local Institution - 0237, Bogotá
  - Local Institution - 0238, Bogotá
  - Local Institution - 0282, Medellín
- Czechia (4):
  - Local Institution - 0112, Hradec Králové
  - Local Institution - 0113, Olomouc
  - Local Institution - 0111, Prague
  - Local Institution - 0232, Příbram
- Finland (2):
  - Local Institution - 0270, Oulu
  - Local Institution - 0271, Turku
- France (15):
  - Local Institution - 0222, Bron, Rhône
  - Local Institution - 0216, Angers
  - Local Institution - 0229, Besançon
  - Local Institution - 0283, Caen
  - Local Institution - 0218, Créteil
  - Local Institution - 0228, Limoges
  - Local Institution - 0215, Marseille
  - Local Institution - 0230, Paris
  - Local Institution - 0227, Pessac
  - Local Institution - 0223, Rennes
  - Local Institution - 0225, Rouen
  - Local Institution - 0217, Saint-Herblain
  - Local Institution - 0221, Saint-Priest-en-Jarez
  - Local Institution - 0224, Strasbourg
  - Local Institution - 0226, Toulon
- Germany (14):
  - Local Institution - 0231, Magdeburg, Saxony-Anhalt
  - Local Institution - 0213, Bad Berka
  - Local Institution - 0208, Berlin
  - Local Institution - 0205, Essen
  - Local Institution - 0210, Frankfurt
  - Local Institution - 0211, Gera
  - Local Institution - 0203, Großhansdorf
  - Local Institution - 0209, Halle
  - Local Institution - 0202, Heidelberg
  - Local Institution - 0214, Hemer
  - Local Institution - 0206, Immenstadt im Allgäu
  - Local Institution - 0204, München
  - Local Institution - 0201, Stuttgart
  - Local Institution - 0212, Wiesbaden
- Greece (4):
  - Local Institution - 0094, Athens, Attikí
  - Local Institution - 0095, Heraklion
  - Local Institution - 0190, Neo Faliro
  - Local Institution - 0101, Thessaloniki
- Hungary (3):
  - Local Institution - 0025, Budapest
  - Local Institution - 0024, Budapest
  - Local Institution - 0026, Mátraháza
- Ireland (4):
  - Local Institution - 0054, Dublin, Dublin
  - Local Institution - 0053, Beaumont
  - Local Institution - 0055, Galway
  - Local Institution - 0100, Limerick
- Israel (5):
  - Local Institution - 0187, Jerusalem
  - Local Institution - 0186, Kfar Saba
  - Local Institution - 0185, Petah Tikva
  - Local Institution - 0184, Tel Litwinsky
  - Local Institution - 0188, Ẕerifin
- Italy (13):
  - Local Institution - 0083, Milan, Lombardy
  - Azienda Ospedaliera Moscati, Avellino
  - Local Institution - 0179, Bergamo
  - IRCCS Azienda Ospedaliero-Universitaria di Bologna, Policlinico di Sant'Orsola, Bologna
  - Local Institution - 0084, Livorno
  - Policlinico G. Martino, Messina
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan
  - Istituto Nazionale Tumori Fondazione Pascale, Napoli
  - Local Institution - 0087, Perugia
  - Ospedale Santa Maria delle Croci, Ravenna
  - Ifo-Istituto Regina Elena, Roma
  - Local Institution - 0089, Roma
  - Local Institution - 0085, Terni
- Japan (35):
  - Local Institution - 0153, Nagoya, Aichi-ken
  - Local Institution - 0152, Nagoya, Aichi-ken
  - Local Institution - 0260, Chiba, Chiba
  - Local Institution - 0148, Kashiwa-shi, Chiba
  - Local Institution - 0159, Matsuyama, Ehime
  - Local Institution - 0160, Fukuoka, Fukuoka
  - Local Institution - 0259, Kurume-shi, Fukuoka
  - Local Institution - 0255, Ota-shi, Gunma
  - Local Institution - 0258, Hiroshima, Hiroshima
  - Local Institution - 0163, Sapporo, Hokkaido
  - Local Institution - 0253, Sapporo, Hokkaido
  - Local Institution - 0252, Akashi-shi, Hyōgo
  - Local Institution - 0156, Kobe, Hyōgo
  - Local Institution - 0146, Kanazawa, Ishikawa-ken
  - Local Institution - 0161, Yokohama, Kanagawa
  - Local Institution - 0150, Yokohama, Kanagawa
  - Local Institution - 0275, Natori-shi, Miyagi
  - Local Institution - 0254, Sendai, Miyagi
  - Local Institution - 0145, Sendai, Miyagi
  - Local Institution - 0164, Niigata, Niigata
  - Local Institution - 0158, Kurashiki-shi, Okayama-ken
  - Local Institution - 0155, Hirakata-shi, Osaka
  - Local Institution - 0154, Osaka, Osaka
  - Local Institution - 0251, Osakasayama-shi, Osaka
  - Local Institution - 0257, Takatsuki-shi, Osaka
  - Local Institution - 0353, Hidaka-shi, Saitama
  - Local Institution - 0256, Kitaadachi-gun, Saitama
  - Local Institution - 0151, Sunto-gun, Shizuoka
  - Local Institution - 0147, Chuo-ku, Tokyo
  - Local Institution - 0149, Koto-ku, Tokyo
  - Local Institution - 0278, Shinjuku-ku, Tokyo
  - Local Institution - 0157, Wakayama, Wakayama
  - Local Institution - 0354, Ube-shi, Yamaguchi
  - Local Institution - 0165, Okayama
  - Local Institution - 0162, Tokyo
- Lebanon (2):
  - Local Institution - 0287, Beirut
  - Local Institution - 0286, Beirut
- Mexico (12):
  - Local Institution - 0197, Guadalajara, Jalisco
  - Local Institution - 0191, Zapopan, Jalisco
  - Local Institution - 0196, Df, Mexico City
  - Local Institution - 0193, Mexico City, Mexico City
  - Local Institution - 0267, Morelia, Michoacán
  - Local Institution - 0277, Monterrey, Nuevo León
  - Local Institution - 0198, Cuautitlán, State of Mexico
  - Local Institution - 0303, Mérida, Yucatán
  - Local Institution - 0192, Chihuahua City
  - Local Institution - 0195, San Luis Potosí City
  - Local Institution - 0236, San Luis Potosí City
  - Local Institution - 0194, Toluca
- Netherlands (5):
  - Local Institution - 0036, Amsterdam
  - Local Institution - 0189, Amsterdam
  - Local Institution - 0169, Breda
  - Local Institution - 0037, Rotterdam
  - Local Institution - 0039, Veldhoven
- Peru (5):
  - Local Institution - 0262, Lima
  - Local Institution - 0263, Lima
  - Local Institution - 0350, Lima
  - Local Institution - 0261, Lima
  - Local Institution - 0351, Lima
- Poland (7):
  - Local Institution - 0060, Bydgoszcz
  - Local Institution - 0058, Gdansk
  - Local Institution - 0063, Gdynia
  - Local Institution - 0072, Gliwice
  - Local Institution - 0057, Lodz
  - Local Institution - 0059, Warsaw
  - Local Institution - 0070, Wroclaw
- Romania (4):
  - Local Institution - 0167, Craiova
  - Local Institution - 0250, Floreşti
  - Local Institution - 0166, Romania
  - Local Institution - 0284, Sector 2
- Russia (7):
  - Local Institution - 0137, Chelyabinsk
  - Local Institution - 0142, Kazan'
  - Local Institution - 0022, Moscow
  - Local Institution - 0028, Saint Petersburg
  - Local Institution - 0049, Saint Petersburg
  - Local Institution - 0027, Saint Petersburg
  - Local Institution - 0143, Ufa
- South Africa (4):
  - Local Institution - 0264, Pretoria, Gauteng
  - Local Institution - 0234, Sandton, Gauteng
  - Local Institution - 0233, Saxonwold, Johannesburg, Gauteng
  - Local Institution - 0305, Vereeniging
- South Korea (5):
  - Local Institution - 0136, Seongnam-si, Kyǒnggi-do
  - Local Institution - 0249, Cheongju-si
  - Local Institution - 0133, Gangnam-gu
  - Local Institution - 0132, Seoul
  - Local Institution - 0135, Seoul
- Spain (6):
  - Local Institution - 0064, Majadahonda, Madrid
  - Local Institution - 0066, Barcelona
  - Local Institution - 0067, Barcelona
  - Local Institution - 0065, Madrid
  - Local Institution - 0069, Seville
  - Local Institution - 0068, Valencia
- Switzerland (4):
  - Local Institution - 0243, Basel
  - Local Institution - 0246, Chur
  - Local Institution - 0244, Lausanne
  - Local Institution - 0245, Winterthur
- Taiwan (5):
  - Local Institution - 0139, Taichung
  - Local Institution - 0138, Taipei
  - Local Institution - 0140, Taipei
  - Local Institution - 0310, Taipei
  - Local Institution - 0141, Taoyuan
- United Kingdom (10):
  - Local Institution - 0266, Middlesbrough, Cleveland
  - Local Institution - 0098, London, Greater London
  - Local Institution - 0099, Southampton, Hampshire
  - Local Institution - 0118, Leicester, Leicestershire
  - Local Institution - 0265, Birmingham
  - Local Institution - 0051, Cambridgeshire
  - Local Institution - 0109, Edinburgh
  - Local Institution - 0097, London
  - Local Institution - 0050, London
  - Local Institution - 0119, Surrey

REFERENCES:
- [Derived] Peters S, Paz-Ares LG, Reck M, Carbone DP, Brahmer JR, Borghaei H, Lu S, O'Byrne KJ, John T, Ciuleanu TE, Schenker M, Bernabe Caro R, Nishio M, Cobo M, Lee JS, Zurawski B, Pluzanski A, Aoyama T, Tschaika M, Devas V, Grootendorst DJ, Ramalingam SS. Long-Term Survival Outcomes With First-Line Nivolumab Plus Ipilimumab-Based Treatment in Patients With Metastatic NSCLC and Tumor Programmed Death-Ligand 1 Lower Than 1%: A Pooled Analysis. J Thorac Oncol. 2025 Jan;20(1):94-108. doi: 10.1016/j.jtho.2024.09.1439. Epub 2024 Oct 4. PMID 39369790
- [Derived] Mason M, Lapuente-Santana O, Halkola AS, Wang W, Mall R, Xiao X, Kaufman J, Fu J, Pfeil J, Banerjee J, Chung V, Chang H, Chasalow SD, Lin HY, Chai R, Yu T, Finotello F, Mirtti T, Mayranpaa MI, Bao J, Verschuren EW, Ahmed EI, Ceccarelli M, Miller LD, Monaco G, Hendrickx WRL, Sherif S, Yang L, Tang M, Gu SS, Zhang W, Zhang Y, Zeng Z, Das Sahu A, Liu Y, Yang W, Bedognetti D, Tang J, Eduati F, Laajala TD, Geese WJ, Guinney J, Szustakowski JD, Vincent BG, Carbone DP. A community challenge to predict clinical outcomes after immune checkpoint blockade in non-small cell lung cancer. J Transl Med. 2024 Feb 21;22(1):190. doi: 10.1186/s12967-023-04705-3. PMID 38383458
- [Derived] Brahmer JR, Lee JS, Ciuleanu TE, Bernabe Caro R, Nishio M, Urban L, Audigier-Valette C, Lupinacci L, Sangha R, Pluzanski A, Burgers J, Mahave M, Ahmed S, Schoenfeld AJ, Paz-Ares LG, Reck M, Borghaei H, O'Byrne KJ, Gupta RG, Bushong J, Li L, Blum SI, Eccles LJ, Ramalingam SS. Five-Year Survival Outcomes With Nivolumab Plus Ipilimumab Versus Chemotherapy as First-Line Treatment for Metastatic Non-Small-Cell Lung Cancer in CheckMate 227. J Clin Oncol. 2023 Feb 20;41(6):1200-1212. doi: 10.1200/JCO.22.01503. Epub 2022 Oct 12. PMID 36223558
- [Derived] Reck M, Ciuleanu TE, Lee JS, Schenker M, Audigier-Valette C, Zurawski B, Linardou H, Otterson GA, Salman P, Nishio M, de la Mora Jimenez E, Lesniewski-Kmak K, Albert I, Ahmed S, Syrigos K, Penrod JR, Yuan Y, Blum SI, Nathan FE, Sun X, Moreno-Koehler A, Taylor F, O'Byrne KJ. First-Line Nivolumab Plus Ipilimumab Versus Chemotherapy in Advanced NSCLC With 1% or Greater Tumor PD-L1 Expression: Patient-Reported Outcomes From CheckMate 227 Part 1. J Thorac Oncol. 2021 Apr;16(4):665-676. doi: 10.1016/j.jtho.2020.12.019. Epub 2021 Jan 21. PMID 33485960
- [Derived] Hellmann MD, Paz-Ares L, Bernabe Caro R, Zurawski B, Kim SW, Carcereny Costa E, Park K, Alexandru A, Lupinacci L, de la Mora Jimenez E, Sakai H, Albert I, Vergnenegre A, Peters S, Syrigos K, Barlesi F, Reck M, Borghaei H, Brahmer JR, O'Byrne KJ, Geese WJ, Bhagavatheeswaran P, Rabindran SK, Kasinathan RS, Nathan FE, Ramalingam SS. Nivolumab plus Ipilimumab in Advanced Non-Small-Cell Lung Cancer. N Engl J Med. 2019 Nov 21;381(21):2020-2031. doi: 10.1056/NEJMoa1910231. Epub 2019 Sep 28. PMID 31562796
- [Derived] Reck M, Schenker M, Lee KH, Provencio M, Nishio M, Lesniewski-Kmak K, Sangha R, Ahmed S, Raimbourg J, Feeney K, Corre R, Franke FA, Richardet E, Penrod JR, Yuan Y, Nathan FE, Bhagavatheeswaran P, DeRosa M, Taylor F, Lawrance R, Brahmer J. Nivolumab plus ipilimumab versus chemotherapy as first-line treatment in advanced non-small-cell lung cancer with high tumour mutational burden: patient-reported outcomes results from the randomised, open-label, phase III CheckMate 227 trial. Eur J Cancer. 2019 Jul;116:137-147. doi: 10.1016/j.ejca.2019.05.008. Epub 2019 Jun 11. PMID 31195357
- [Derived] Hellmann MD, Ciuleanu TE, Pluzanski A, Lee JS, Otterson GA, Audigier-Valette C, Minenza E, Linardou H, Burgers S, Salman P, Borghaei H, Ramalingam SS, Brahmer J, Reck M, O'Byrne KJ, Geese WJ, Green G, Chang H, Szustakowski J, Bhagavatheeswaran P, Healey D, Fu Y, Nathan F, Paz-Ares L. Nivolumab plus Ipilimumab in Lung Cancer with a High Tumor Mutational Burden. N Engl J Med. 2018 May 31;378(22):2093-2104. doi: 10.1056/NEJMoa1801946. Epub 2018 Apr 16. PMID 29658845
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.BMSClinicalTrials.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Part 1-Arm B: Nivo + Ipi: Participants with PD-L1 positive status Non Small Cell Lung Cancer received nivolumab 3 mg/kg IV over 30 minutes Q2W + ipilimumab 1 mg/kg over 30minutes every 6 weeks (Q6W) given for up to 24 months in the absence of disease progression or unacceptable toxicity.
- Part 1-Arm A: Nivolumab: Participants with PD-L1 positive status Non Small Cell Lung Cancer received nivolumab 240 mg intravenously (IV) over 30 minutes every 2 weeks (Q2W) given for up to 24months in the absence of disease progression or unacceptable toxicity.
- Part 1-Arm C: Chemotherapy: Participants with PD-L1 positive status Non Small Cell Lung Cancer received histology-based platinum-doublet chemotherapy IV in3-week cycles for a maximum of 4 cycles or until disease progression or unacceptable toxicity (whichever comes first). For participants with NSQ histology, pemetrexed maintenance was allowed until disease progression or unacceptable toxicity after 4 cycles of chemotherapy.
- Part 1-Arm D: Nivo + Ipi: Participants with PD-L1 negative status Non Small Cell Lung Cancer received nivolumab 3 mg/kg IV over 30 minutes Q2W + ipilimumab 1 mg/kg over 30minutes Q6W given for up to 24 months in the absence of disease progression or unacceptable toxicity.
- Part 1-Arm G: Nivo + Chemo: Participants with PD-L1 negative status Non Small Cell Lung Cancer received nivolumab 360 mg IV over 30 minutes combined with platinum-doublet chemotherapy administered IV every 3 weeks for a maximum of 4 cycles. Participants who have not experienced disease progression were to receive nivolumab 360 mg every 3weeks until the progression of disease, discontinuation due to toxicity, or up to 24 months (whichever comes first). For subjects with NSQ histology, pemetrexed maintenance was allowed until disease progression or unacceptable toxicity after 4 cycles of chemotherapy.
- Part 1-Arm F: Chemotherapy: Participants with PD-L1 negative status Non Small Cell Lung Cancer received histology-based platinum-doublet chemotherapy IV in 3-week cycles for a maximum of 4 cycles or until disease progression or unacceptable toxicity (whichever comes first). For participants with NSQ histology, pemetrexed maintenance was allowed until disease progression or unacceptable toxicity after 4 cycles of chemotherapy.
- Part 2 - Arm H: Nivolumab + Chemotherapy: Chemotherapy-naive participants with stage IV or recurrent NSCLC irrespective of PD-L1 expressing levels received nivolumab 360 mg IV over 30 minutes combined with platinum-doublet chemotherapy administered IV every 3 weeks for a maximum of 4 cycles. Participants who have not experienced disease progression were to receive nivolumab 360 mg every 3weeks until the progression of disease, discontinuation due to toxicity, or up to 24 months (whichever comes first). For subjects with NSQ histology, pemetrexed maintenance was allowed until disease progression or unacceptable toxicity after 4 cycles of chemotherapy.
- Part 2 - Arm I: Chemotherapy: Chemotherapy-naive participants with stage IV or recurrent NSCLC irrespective of PD-L1 expressing levels received histology-based platinum-doublet chemotherapy IV in 3-week cycles for a maximum of 4 cycles or until disease progression or unacceptable toxicity (whichever comes first). For participants with NSQ histology, pemetrexed maintenance was allowed until disease progression or unacceptable toxicity after 4 cycles of chemotherapy.
- Part 3 -Arm J: Nivolumab + Ipilimumab: Participants in China with PD-L1 Non Small Cell Lung Cancer received nivolumab 3 mg/kg IV over 30 minutes Q2W + ipilimumab 1 mg/kg over 30minutes every 6 weeks (Q6W) given for up to 24 months in the absence of disease progression or unacceptable toxicity.
- Part 3 - Arm K: Chemotherapy: Participants in China with PD-L1 Non Small Cell Lung Cancer received histology-based platinum-doublet chemotherapy IV in3-week cycles for a maximum of 4 cycles or until disease progression or unacceptable toxicity (whichever comes first). For participants with NSQ histology, pemetrexed maintenance was allowed until disease progression or unacceptable toxicity after 4 cycles of chemotherapy.
Period: Pre-Treatment
Arm/Group | Part 1-Arm B: Nivo + Ipi | Part 1-Arm A: Nivolumab | Part 1-Arm C: Chemotherapy | Part 1-Arm D: Nivo + Ipi | Part 1-Arm G: Nivo + Chemo | Part 1-Arm F: Chemotherapy | Part 2 - Arm H: Nivolumab + Chemotherapy | Part 2 - Arm I: Chemotherapy | Part 3 -Arm J: Nivolumab + Ipilimumab | Part 3 - Arm K: Chemotherapy
Started | 396 | 396 | 397 | 187 | 177 | 186 | 377 | 378 | 126 | 127
Completed | 391 | 391 | 387 | 185 | 172 | 183 | 375 | 371 | 126 | 123
Not Completed | 5 | 5 | 10 | 2 | 5 | 3 | 2 | 7 | 0 | 4
Not completed — Adverse events unrelated to study drug | 0 | 1 | 2 | 1 | 0 | 0 | 1 | 5 | 0 | 0
Not completed — Other reasons | 4 | 1 | 4 | 1 | 4 | 2 | 0 | 0 | 0 | 0
Not completed — Subject no longer meets study criteria | 1 | 2 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Not completed — Subject withdrew consent | 0 | 0 | 3 | 0 | 0 | 1 | 0 | 1 | 0 | 3
Not completed — Subject request to discontinue study treatment | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Period: Treatment Period
Arm/Group | Part 1-Arm B: Nivo + Ipi | Part 1-Arm A: Nivolumab | Part 1-Arm C: Chemotherapy | Part 1-Arm D: Nivo + Ipi | Part 1-Arm G: Nivo + Chemo | Part 1-Arm F: Chemotherapy | Part 2 - Arm H: Nivolumab + Chemotherapy | Part 2 - Arm I: Chemotherapy | Part 3 -Arm J: Nivolumab + Ipilimumab | Part 3 - Arm K: Chemotherapy
Started | 391 | 391 | 387 | 185 | 172 | 183 | 375 | 371 | 126 | 123
Completed | 45 | 37 | 94 | 14 | 20 | 32 | 40 | 83 | 0 | 37
Not Completed | 346 | 354 | 293 | 171 | 152 | 151 | 335 | 288 | 126 | 86
Not completed — Not reported | 8 | 6 | 4 | 4 | 2 | 1 | 14 | 8 | 5 | 2
Not completed — Other reasons | 5 | 6 | 12 | 7 | 5 | 1 | 8 | 8 | 21 | 1
Not completed — Administrative reason by sponsor | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Participant meet no longer study criteria | 1 | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0
Not completed — Poor/Non Compliance | 1 | 0 | 2 | 0 | 0 | 1 | 1 | 0 | 0 | 1
Not completed — Maximum Clinical Benefit | 3 | 3 | 1 | 1 | 3 | 0 | 3 | 2 | 2 | 2
Not completed — Lost to Follow-up | 0 | 0 | 1 | 1 | 0 | 0 | 2 | 2 | 0 | 0
Not completed — Participant withdrew Consent | 5 | 5 | 3 | 3 | 1 | 3 | 3 | 3 | 2 | 3
Not completed — Participant request to discontinue treatment | 5 | 3 | 15 | 5 | 3 | 6 | 13 | 15 | 4 | 18
Not completed — Adverse event unrelated to study drug | 23 | 29 | 22 | 18 | 11 | 15 | 25 | 19 | 4 | 2
Not completed — Death | 4 | 7 | 0 | 0 | 1 | 2 | 6 | 5 | 9 | 0
Not completed — Study Drug Toxicity | 79 | 51 | 31 | 39 | 12 | 25 | 52 | 30 | 20 | 9
Not completed — Disease progression | 212 | 240 | 202 | 93 | 113 | 96 | 208 | 195 | 59 | 46
Not completed — Pregnancy | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Other | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1-Arm B: Nivo + Ipi | Part 1-Arm A: Nivolumab | Part 1-Arm C: Chemotherapy | Part 1-Arm D: Nivo + Ipi | Part 1-Arm G: Nivo + Chemo | Part 1-Arm F: Chemotherapy | Part 2 - Arm H: Nivolumab + Chemotherapy | Part 2 - Arm I: Chemotherapy | Part 3 -Arm J: Nivolumab + Ipilimumab | Part 3 - Arm K: Chemotherapy | Total
Number analyzed (Participants) | 396 | 396 | 397 | 187 | 177 | 186 | 377 | 378 | 126 | 127 | 2747
Age, Customized [Count of Participants; unit: Participants]
  < 65 | 199 | 210 | 207 | 107 | 91 | 98 | 214 | 196 | 82 | 84 | 1488
  =>65 | 197 | 186 | 190 | 80 | 86 | 88 | 163 | 182 | 44 | 43 | 1259
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 141 | 124 | 137 | 49 | 47 | 61 | 113 | 115 | 18 | 20 | 825
  Male | 255 | 272 | 260 | 138 | 130 | 125 | 264 | 263 | 108 | 107 | 1922
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 299 | 317 | 305 | 143 | 136 | 133 | 272 | 266 | 0 | 0 | 1871
  Black | 4 | 6 | 5 | 0 | 2 | 2 | 1 | 3 | 0 | 0 | 23
  Asian | 84 | 67 | 82 | 41 | 38 | 45 | 93 | 94 | 126 | 127 | 797
  Other | 5 | 6 | 3 | 1 | 1 | 5 | 8 | 12 | 0 | 0 | 41
  American Indian or Alaska Native | 4 | 0 | 2 | 2 | 0 | 1 | 3 | 1 | 0 | 0 | 13
  Native Hawaiian or other pacific islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival Per BICR
Description: Progression-Free Survival then (PFS) is defined as the time between the date of randomization and the date of first documented disease progression, based on BICR assessments (per RECIST v1.1), or death due to any cause, whichever occurs first based on Kaplan-Meier estimates. Progressive Disease (PD): At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum during the study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm.
Time Frame: From randomization untill disease progression or death, whichever occurs first (up to approximately 481 weeks)
Population: All randomized participants
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Part 1-Arm B: Nivo + Ipi | Part 1-Arm A: Nivolumab | Part 1-Arm C: Chemotherapy | Part 1-Arm D: Nivo + Ipi | Part 1-Arm G: Nivo + Chemo | Part 1-Arm F: Chemotherapy | Part 2 - Arm H: Nivolumab + Chemotherapy | Part 2 - Arm I: Chemotherapy | Part 3 -Arm J: Nivolumab + Ipilimumab | Part 3 - Arm K: Chemotherapy
Number analyzed (Participants) | 396 | 396 | 397 | 187 | 177 | 186 | 377 | 378 | 126 | 127
months | 5.06 [4.07 to 6.31] | 4.17 [3.22 to 5.32] | 5.55 [4.63 to 5.82] | 4.90 [3.15 to 6.28] | 5.55 [4.63 to 6.90] | 4.70 [4.21 to 5.59] | 8.34 [7.10 to 9.59] | 5.52 [4.47 to 5.85] | 5.78 [4.14 to 8.34] | 5.49 [4.37 to 6.77]
Statistical Analysis 1: Comparison: Part 1-Arm B: Nivo + Ipi vs Part 1-Arm C: Chemotherapy; Test type: Superiority; Hazard Ratio (HR) = 0.79, 95% CI 2-sided [0.67 to 0.93]
Statistical Analysis 2: Comparison: Part 1-Arm A: Nivolumab vs Part 1-Arm C: Chemotherapy; Test type: Superiority; Hazard Ratio (HR) = 0.95, 95% CI 2-sided [0.81 to 1.12]
Statistical Analysis 3: Comparison: Part 1-Arm B: Nivo + Ipi vs Part 1-Arm A: Nivolumab; Test type: Superiority; Hazard Ratio (HR) = 0.85, 95% CI 2-sided [0.72 to 0.99]
Statistical Analysis 4: Comparison: Part 1-Arm D: Nivo + Ipi vs Part 1-Arm F: Chemotherapy; Test type: Superiority; Cox Proportional Hazard = 0.76, 95% CI 2-sided [0.60 to 0.97]
Statistical Analysis 5: Comparison: Part 1-Arm G: Nivo + Chemo vs Part 1-Arm F: Chemotherapy; Test type: Superiority; Hazard Ratio (HR) = 0.74, 95% CI 2-sided [0.59 to 0.93]
Statistical Analysis 6: Comparison: Part 2 - Arm H: Nivolumab + Chemotherapy vs Part 2 - Arm I: Chemotherapy; Test type: Superiority; Hazard Ratio (HR) = 0.61, 95% CI 2-sided [0.52 to 0.72]
Statistical Analysis 7: Comparison: Part 3 -Arm J: Nivolumab + Ipilimumab vs Part 3 - Arm K: Chemotherapy; Test type: Superiority; Hazard Ratio (HR) = 0.66, 95% CI 2-sided [0.49 to 0.89]

2. Primary Outcome: Overall Survival
Description: OS for all randomized participants is the time between randomization date and the date of death from any cause.
Time Frame: From randomization untill death or last follow up whichever occurs first (up to approximately 481 weeks)
Population: All randomized participants
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Part 1-Arm B: Nivo + Ipi | Part 1-Arm A: Nivolumab | Part 1-Arm C: Chemotherapy | Part 1-Arm D: Nivo + Ipi | Part 1-Arm G: Nivo + Chemo | Part 1-Arm F: Chemotherapy | Part 2 - Arm H: Nivolumab + Chemotherapy | Part 2 - Arm I: Chemotherapy | Part 3 -Arm J: Nivolumab + Ipilimumab | Part 3 - Arm K: Chemotherapy
Number analyzed (Participants) | 396 | 396 | 397 | 187 | 177 | 186 | 377 | 378 | 126 | 127
months | 17.12 [14.95 to 20.17] | 15.70 [13.27 to 18.14] | 14.88 [12.71 to 16.72] | 17.45 [13.21 to 22.05] | 15.21 [12.29 to 19.78] | 12.19 [9.17 to 14.32] | 18.27 [15.84 to 21.65] | 14.72 [12.42 to 16.79] | 20.99 [16.95 to 25.17] | 15.11 [13.17 to 18.89]
Statistical Analysis 1: Comparison: Part 1-Arm B: Nivo + Ipi vs Part 1-Arm C: Chemotherapy; Test type: Superiority; Hazard Ratio (HR) = 0.78, 95% CI 2-sided [0.67 to 0.91]
Statistical Analysis 2: Comparison: Part 1-Arm A: Nivolumab vs Part 1-Arm C: Chemotherapy; Test type: Superiority; Hazard Ratio (HR) = 0.91, 95% CI 2-sided [0.78 to 1.05]
Statistical Analysis 3: Comparison: Part 1-Arm B: Nivo + Ipi vs Part 1-Arm A: Nivolumab; Test type: Superiority; Hazard Ratio (HR) = 0.86, 95% CI 2-sided [0.74 to 1.01]
Statistical Analysis 4: Comparison: Part 1-Arm D: Nivo + Ipi vs Part 1-Arm F: Chemotherapy; Test type: Superiority; Hazard Ratio (HR) = 0.64, 95% CI 2-sided [0.51 to 0.79]
Statistical Analysis 5: Comparison: Part 1-Arm G: Nivo + Chemo vs Part 1-Arm F: Chemotherapy; Test type: Superiority; Hazard Ratio (HR) = 0.77, 95% CI 2-sided [0.63 to 0.96]
Statistical Analysis 6: Comparison: Part 2 - Arm H: Nivolumab + Chemotherapy vs Part 2 - Arm I: Chemotherapy; Test type: Superiority; Hazard Ratio (HR) = 0.75, 95% CI 2-sided [0.64 to 0.87]
Statistical Analysis 7: Comparison: Part 3 -Arm J: Nivolumab + Ipilimumab vs Part 3 - Arm K: Chemotherapy; Test type: Superiority; Hazard Ratio (HR) = 0.85, 95% CI 2-sided [0.64 to 1.14]

3. Secondary Outcome: Objective Response Rate (ORR) Per BICR
Description: Objective response rate (ORR) is defined as the number of participants who achieve a best overall response (BOR) of confirmed complete response (CR) or confirmed partial response (PR), based on blinded independent central review (BICR) assessments using Response Evaluation Criteria in Solid Tumors (RECIST 1.1), divided by the number of all randomized participants.
  Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm.
  Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: From randomization untill disease progression or death, whichever occurs first (up to approximately 481 weeks)
Population: All randomized participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 1-Arm B: Nivo + Ipi | Part 1-Arm A: Nivolumab | Part 1-Arm C: Chemotherapy | Part 1-Arm D: Nivo + Ipi | Part 1-Arm G: Nivo + Chemo | Part 1-Arm F: Chemotherapy | Part 2 - Arm H: Nivolumab + Chemotherapy | Part 2 - Arm I: Chemotherapy | Part 3 -Arm J: Nivolumab + Ipilimumab | Part 3 - Arm K: Chemotherapy
Number analyzed (Participants) | 396 | 396 | 397 | 187 | 177 | 186 | 377 | 378 | 126 | 127
percentage of participants | 36.4 [31.6 to 41.3] | 27.5 [23.2 to 32.2] | 29.7 [25.3 to 34.5] | 26.2 [20.1 to 33.1] | 37.9 [30.7 to 45.4] | 23.1 [17.3 to 29.8] | 52.3 [47.1 to 57.4] | 29.9 [25.3 to 34.8] | 38.1 [29.6 to 47.2] | 30.7 [22.8 to 39.5]

4. Secondary Outcome: Percentage of Participants With Symptom Deterioration at Week 12 Assessed Via Lung Cancer Symptom Scale
Description: The Lung Cancer Symptom Scale (LCSS) is a disease measure of quality of life which evaluates six major lung cancer symptoms and their effect on overall distress and symptom severity, impact on day-to-day activities, and overall quality of life. This patient reported outcome (PRO) questionnaire assesses the following 6 symptoms items (appetite loss, fatigue, cough, dyspnea, hemoptysis, pain) and 3 summary global items (symptom distress, activity level, overall quality of life) for patients using visual analogue scales (VAS) (100 mm horizontal line) ranging from 0 (best rating) to 100 (worst rating). The LCSS average total score is sum of items 1 to 9 divided by the total number of items ((sum of items 1 to 9)/9) ranging from 0 to 100 where high score represent worst outcome. Disease-Related Symptom Deterioration by Week 12 defined as a 10 points or more increase from baseline in LCSS average score at any time (on or off-treatment) up to 95 days from randomization date.
Time Frame: Week 12
Population: All randomized participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 1-Arm B: Nivo + Ipi | Part 1-Arm A: Nivolumab | Part 1-Arm C: Chemotherapy | Part 1-Arm D: Nivo + Ipi | Part 1-Arm G: Nivo + Chemo | Part 1-Arm F: Chemotherapy | Part 2 - Arm H: Nivolumab + Chemotherapy | Part 2 - Arm I: Chemotherapy | Part 3 -Arm J: Nivolumab + Ipilimumab | Part 3 - Arm K: Chemotherapy
Number analyzed (Participants) | 396 | 396 | 397 | 187 | 177 | 186 | 377 | 378 | 126 | 127
percentage of participants | 31.3 [26.8 to 36.1] | 35.4 [30.6 to 40.3] | 25.7 [21.5 to 30.3] | 33.2 [26.5 to 40.4] | 28.8 [22.3 to 36.1] | 37.6 [30.7 to 45.0] | 30.0 [25.4 to 34.9] | 24.3 [20.1 to 29.0] | 23.0 [16.0 to 31.4] | 26.0 [18.6 to 34.5]

ADVERSE EVENTS:
Time Frame: Serious and non-serious adverse events were collected from first dose (Day 1) and 30 days after last dose of study therapy (up to approximately 105 months) and all cause mortality was collected from Day 1 and up to 481 weeks.
Description: Randomized participants
Arm/Group | Part 1-Arm B: Nivo + Ipi | Part 1-Arm A: Nivolumab | Part 1-Arm C: Chemotherapy | Part 1-Arm D: Nivo + Ipi | Part 1-Arm G: Nivo + Chemo | Part 1-Arm F: Chemotherapy | Part 2 - Arm H: Nivolumab + Chemotherapy | Part 2 - Arm I: Chemotherapy | Part 3 -Arm J: Nivolumab + Ipilimumab | Part 3 - Arm K: Chemotherapy
All-Cause Mortality (participants affected / at risk) | 316/391 | 333/391 | 339/387 | 159/185 | 157/172 | 174/183 | 314/375 | 335/371 | 95/126 | 94/123
Serious Adverse Events (participants affected / at risk) | 275/391 | 239/391 | 213/387 | 128/185 | 112/172 | 91/183 | 240/375 | 180/371 | 78/126 | 60/123
Other Adverse Events (participants affected / at risk) | 366/391 | 356/391 | 361/387 | 172/185 | 167/172 | 165/183 | 357/375 | 345/371 | 124/126 | 121/123
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1-Arm B: Nivo + Ipi (N=391) | Part 1-Arm A: Nivolumab (N=391) | Part 1-Arm C: Chemotherapy (N=387) | Part 1-Arm D: Nivo + Ipi (N=185) | Part 1-Arm G: Nivo + Chemo (N=172) | Part 1-Arm F: Chemotherapy (N=183) | Part 2 - Arm H: Nivolumab + Chemotherapy (N=375) | Part 2 - Arm I: Chemotherapy (N=371) | Part 3 -Arm J: Nivolumab + Ipilimumab (N=126) | Part 3 - Arm K: Chemotherapy (N=123)
Anaemia (Blood and lymphatic system disorders) | 4 | 4 | 9 | 4 | 10 | 8 | 14 | 10 | 1 | 2
Autoimmune haemolytic anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bone marrow failure (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Eosinophilia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Febrile bone marrow aplasia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 3 | 9 | 2 | 4 | 7 | 16 | 6 | 0 | 0
Haematotoxicity (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Heparin-induced thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Myelosuppression (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 7
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 2 | 0 | 1 | 0 | 1 | 1 | 0 | 1
Pancytopenia (Blood and lymphatic system disorders) | 0 | 3 | 2 | 0 | 4 | 1 | 5 | 4 | 0 | 0
Splenic haematoma (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Splenic haemorrhage (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Splenic thrombosis (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 5 | 0 | 4 | 1 | 2 | 2 | 0 | 2
Thrombocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Acute coronary syndrome (Cardiac disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute left ventricular failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 2 | 1 | 0 | 2 | 0 | 0 | 2 | 0 | 0 | 0
Angina pectoris (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Angina unstable (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Arrhythmia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Arteriosclerosis coronary artery (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 4 | 4 | 0 | 4 | 1 | 0 | 3 | 0 | 0 | 0
Atrial flutter (Cardiac disorders) | 1 | 1 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Atrioventricular block complete (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac arrest (Cardiac disorders) | 2 | 4 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cardiac failure (Cardiac disorders) | 3 | 2 | 1 | 3 | 1 | 2 | 2 | 0 | 0 | 0
Cardiac failure acute (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 2 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Cardiac fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cardiac tamponade (Cardiac disorders) | 1 | 3 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Cardio-respiratory arrest (Cardiac disorders) | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 1 | 0
Cardiogenic shock (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cardiopulmonary failure (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Coronary artery disease (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 1
Hypertensive cardiomyopathy (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Immune-mediated myocarditis (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Myocardial infarction (Cardiac disorders) | 2 | 0 | 1 | 3 | 1 | 0 | 1 | 0 | 0 | 0
Myocardial ischaemia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Myocarditis (Cardiac disorders) | 2 | 0 | 0 | 0 | 1 | 0 | 3 | 1 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pericardial effusion (Cardiac disorders) | 2 | 5 | 2 | 1 | 1 | 1 | 0 | 3 | 2 | 1
Pericardial effusion malignant (Cardiac disorders) | 0 | 4 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0
Pericarditis (Cardiac disorders) | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Pleuropericarditis (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Right ventricular failure (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Stress cardiomyopathy (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Supraventricular extrasystoles (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Supraventricular tachyarrhythmia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Torsade de pointes (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tracheo-oesophageal fistula (Congenital, familial and genetic disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sudden hearing loss (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Adrenal insufficiency (Endocrine disorders) | 10 | 1 | 0 | 6 | 1 | 0 | 1 | 0 | 0 | 0
Autoimmune hypothyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Autoimmune thyroiditis (Endocrine disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypercalcaemia of malignancy (Endocrine disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperparathyroidism secondary (Endocrine disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperthyroidism (Endocrine disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypophysitis (Endocrine disorders) | 5 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 2 | 0
Hypopituitarism (Endocrine disorders) | 5 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypothyroidism (Endocrine disorders) | 1 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Immune-mediated hypophysitis (Endocrine disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Primary adrenal insufficiency (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Secondary adrenocortical insufficiency (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cataract (Eye disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Diplopia (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal hernia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 2 | 2 | 0 | 1 | 0 | 4 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Autoimmune colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 9 | 4 | 0 | 3 | 1 | 0 | 4 | 1 | 0 | 0
Colitis ischaemic (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Colitis microscopic (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Colitis ulcerative (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 3 | 2 | 2 | 2 | 0 | 3 | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 6 | 3 | 4 | 9 | 1 | 3 | 6 | 2 | 4 | 2
Duodenal ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 3 | 1 | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 0
Enterocolitis (Gastrointestinal disorders) | 3 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Erosive oesophagitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 3 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gingival hypertrophy (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ileus (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Immune-mediated enterocolitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Immune-mediated gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Immune-mediated pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Intestinal ischaemia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Large intestinal ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Large intestine perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Malignant ascites (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Melaena (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 2 | 7 | 1 | 1 | 4 | 2 | 4 | 1 | 0
Odynophagia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oesophageal fistula (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Oesophageal stenosis (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oesophageal ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Oesophagitis (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0
Rectal ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Subileus (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 7 | 7 | 2 | 1 | 2 | 5 | 4 | 1 | 0
Adverse drug reaction (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Asthenia (General disorders) | 3 | 4 | 5 | 5 | 2 | 0 | 2 | 3 | 0 | 0
Chest discomfort (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Chest pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Chills (General disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Complication associated with device (General disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Death (General disorders) | 1 | 2 | 1 | 1 | 0 | 3 | 1 | 1 | 1 | 1
Drug withdrawal syndrome (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Face oedema (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 3 | 3 | 1 | 1 | 4 | 1 | 1 | 2 | 0 | 0
General physical health deterioration (General disorders) | 0 | 4 | 3 | 1 | 1 | 4 | 1 | 3 | 0 | 0
Generalised oedema (General disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperthermia (General disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypothermia (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Inflammation (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Influenza like illness (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Malaise (General disorders) | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Mucosal inflammation (General disorders) | 0 | 3 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Multiple organ dysfunction syndrome (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 1 | 1 | 0 | 1 | 1 | 3 | 0 | 0 | 0
Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Performance status decreased (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 5 | 5 | 5 | 3 | 3 | 3 | 6 | 5 | 6 | 0
Sudden death (General disorders) | 3 | 5 | 0 | 0 | 1 | 1 | 6 | 2 | 4 | 1
Swelling (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Systemic inflammatory response syndrome (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Acute hepatic failure (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Autoimmune hepatitis (Hepatobiliary disorders) | 3 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 1 | 0
Bile duct stone (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Biliary obstruction (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cholangitis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cholangitis acute (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 2 | 1 | 0 | 0 | 1 | 2 | 0 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cholestasis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 3
Hepatic failure (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 2 | 0 | 0 | 2 | 0 | 1 | 1 | 0 | 0 | 0
Hepatitis (Hepatobiliary disorders) | 3 | 4 | 0 | 6 | 0 | 0 | 0 | 0 | 1 | 0
Hepatorenal failure (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hepatotoxicity (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hydrocholecystis (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypertransaminasaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Immune-mediated hepatic disorder (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Immune-mediated hepatitis (Hepatobiliary disorders) | 3 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 7 | 0
Jaundice cholestatic (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Liver disorder (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Liver injury (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Anaphylactic reaction (Immune system disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Anaphylactic shock (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Contrast media allergy (Immune system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Contrast media reaction (Immune system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Infusion related hypersensitivity reaction (Immune system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abscess limb (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Anal abscess (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 4 | 0 | 1 | 0
Aspergillus infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Bacterial diarrhoea (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Bacterial infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 3 | 1 | 1 | 1 | 1 | 0 | 5 | 0 | 0 | 0
Bronchopulmonary aspergillosis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Catheter site infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 1 | 0 | 4 | 0 | 3 | 4 | 0 | 0
Clostridium difficile infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dermo-hypodermitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Diabetic foot infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diverticulitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0
Diverticulitis intestinal perforated (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Empyema (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Encephalitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Enteritis infectious (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Enterocolitis infectious (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Erysipelas (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Febrile infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 1 | 1 | 0 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Groin infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Infection (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Infectious pleural effusion (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Injection site infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Klebsiella urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Large intestine infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 1 | 1 | 1 | 3 | 0 | 2 | 2 | 0 | 0
Lung abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Meningitis viral (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Metapneumovirus infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myelitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neutropenic infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Neutropenic sepsis (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 1 | 2 | 0 | 0 | 0
Oesophageal candidiasis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ophthalmic herpes zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Osteomyelitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Parainfluenzae virus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Peritonitis (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0
Pleural infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 40 | 29 | 31 | 18 | 15 | 8 | 34 | 29 | 11 | 8
Pneumonia adenoviral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pneumonia aspiration (Infections and infestations) | 1 | 2 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0
Pneumonia bacterial (Infections and infestations) | 1 | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 0
Pneumonia influenzal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pneumonia klebsiella (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia necrotising (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pneumonia viral (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Pseudomembranous colitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary sepsis (Infections and infestations) | 1 | 3 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary tuberculosis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyelonephritis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rectal abscess (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory syncytial virus infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 4 | 5 | 3 | 4 | 2 | 1 | 1 | 3 | 1 | 0
Respiratory tract infection viral (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Salmonellosis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 3 | 3 | 3 | 1 | 1 | 4 | 7 | 2 | 0 | 0
Septic shock (Infections and infestations) | 2 | 4 | 1 | 4 | 0 | 2 | 1 | 1 | 1 | 0
Skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Soft tissue infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Staphylococcal infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Systemic candida (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Thrombophlebitis septic (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tooth infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 5 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 4 | 2 | 4 | 1 | 1 | 0 | 2 | 3 | 0 | 1
Urosepsis (Infections and infestations) | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 2 | 0 | 0
Vascular device infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Viral infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Viral pericarditis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Wound infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Accidental overdose (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Acetabulum fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Femoral nerve injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 3 | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 0
Forearm fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Fracture displacement (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 1 | 2 | 1 | 0 | 0 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Multiple fractures (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscle strain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Post procedural complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Radiation oesophagitis (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Radiation pneumonitis (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 2 | 3 | 0 | 1 | 2 | 0 | 0 | 1 | 1 | 0
Amylase increased (Investigations) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood calcium decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blood creatinine increased (Investigations) | 1 | 0 | 1 | 0 | 0 | 0 | 3 | 0 | 0 | 0
Blood glucose increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood potassium decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eosinophil count increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
General physical condition abnormal (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hepatic enzyme increased (Investigations) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lipase increased (Investigations) | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Liver function test abnormal (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Liver function test increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lymphocyte count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 3 | 0 | 4
Pancreatic enzymes increased (Investigations) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Platelet count decreased (Investigations) | 0 | 0 | 3 | 0 | 0 | 1 | 6 | 2 | 3 | 8
Transaminases increased (Investigations) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Troponin increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Weight decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 2
Acidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Adult failure to thrive (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 2 | 0 | 1 | 0 | 1 | 4 | 3 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 4 | 1 | 0 | 1 | 1 | 1 | 1 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Diabetic metabolic decompensation (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Failure to thrive (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 3 | 4 | 1 | 1 | 0 | 0 | 0 | 2 | 0 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 0 | 1 | 3 | 0 | 0 | 4 | 1 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 1 | 0 | 1 | 1 | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 3 | 3 | 2 | 1 | 1 | 0 | 6 | 1 | 3 | 0
Hypoproteinaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ketoacidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 3 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 2 | 0 | 1 | 0
Autoimmune arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 1 | 3 | 1 | 0 | 2 | 0 | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypertrophic osteoarthropathy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Myopathy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Myositis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Polyarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Benign breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 3 | 3 | 3 | 1 | 1 | 1 | 5 | 1 | 1
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Extranodal marginal zone B-cell lymphoma (MALT type) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Female reproductive neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gastric neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Haematological malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hepatobiliary cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Infected neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Intestinal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Intestinal metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lymphangiosis carcinomatosa (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 98 | 102 | 87 | 39 | 48 | 41 | 81 | 78 | 18 | 9
Metastases to adrenals (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 0 | 0
Metastases to pleura (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oncologic complication (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Paraneoplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Tumour compression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tumour invasion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tumour necrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2 | 1 | 0 | 0 | 0 | 2 | 1 | 1 | 0
Tumour pseudoprogression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Atonic seizures (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Brain oedema (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Cerebellar infarction (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cerebral infarction (Nervous system disorders) | 0 | 1 | 4 | 1 | 1 | 0 | 0 | 1 | 0 | 0
Cerebral ischaemia (Nervous system disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cerebral microangiopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 4 | 5 | 3 | 3 | 2 | 1 | 1 | 3 | 0 | 0
Cerebrovascular disorder (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 2 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Dysarthria (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Embolic cerebral infarction (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Encephalitis autoimmune (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Encephalopathy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Epilepsy (Nervous system disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0
Facial paralysis (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Generalised tonic-clonic seizure (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemorrhage intracranial (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Haemorrhagic cerebral infarction (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Haemorrhagic stroke (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemorrhagic transformation stroke (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hemiparesis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 1 | 3 | 2 | 0 | 0 | 1 | 1 | 0 | 0
Lethargy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lumbar radiculopathy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myasthenia gravis (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Myasthenic syndrome (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nerve compression (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Neuralgia (Nervous system disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Paralysis recurrent laryngeal nerve (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Paraplegia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Partial seizures (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Polyneuropathy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Quadriparesis (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Seizure (Nervous system disorders) | 2 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Sensory loss (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Spinal cord compression (Nervous system disorders) | 0 | 0 | 2 | 0 | 1 | 1 | 0 | 1 | 0 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 2 | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vasogenic cerebral oedema (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vertebrobasilar artery dissection (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vocal cord paralysis (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Device dislocation (Product Issues) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Device physical property issue (Product Issues) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Bipolar disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Completed suicide (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Confusional state (Psychiatric disorders) | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Delirium (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Disorientation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Mental status changes (Psychiatric disorders) | 0 | 2 | 1 | 0 | 2 | 0 | 2 | 0 | 0 | 0
Suicide attempt (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 2 | 4 | 4 | 3 | 2 | 0 | 2 | 2 | 0 | 1
Autoimmune nephritis (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Azotaemia (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nephrogenic diabetes insipidus (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nephropathy toxic (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 3 | 1 | 2 | 0 | 1 | 0 | 3 | 3 | 1 | 0
Renal vascular thrombosis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tubulointerstitial nephritis (Renal and urinary disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ureterolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Intermenstrual bleeding (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ovarian cyst (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vaginal prolapse (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Apnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0
Bronchial haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 1 | 2 | 5 | 1 | 0 | 1 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8 | 9 | 8 | 2 | 1 | 2 | 4 | 5 | 1 | 1
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 7 | 3 | 0 | 0 | 2 | 1 | 4 | 1
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Immune-mediated lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 4 | 2 | 1 | 2 | 1 | 0 | 1 | 0 | 3 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lung opacity (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Malignant pleural effusion (Respiratory, thoracic and mediastinal disorders) | 9 | 4 | 1 | 3 | 1 | 4 | 2 | 2 | 0 | 0
Mediastinal disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Oesophagobronchial fistula (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 5 | 4 | 1 | 1 | 3 | 1 | 7 | 5 | 3 | 1
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 20 | 11 | 4 | 7 | 5 | 1 | 14 | 1 | 11 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 2 | 1 | 0 | 1 | 5 | 1 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 13 | 7 | 5 | 4 | 6 | 2 | 9 | 5 | 0 | 1
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pulmonary hilum mass (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary venous thrombosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory alkalosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 4 | 5 | 5 | 3 | 3 | 6 | 3 | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Autoimmune dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diabetic foot (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Exfoliative rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neutrophilic dermatosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash vesicular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aortic thrombosis (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arterial thrombosis (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arteritis (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Circulatory collapse (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 2 | 2 | 2 | 2 | 0 | 1 | 4 | 0 | 0 | 0
Embolism (Vascular disorders) | 2 | 3 | 2 | 0 | 0 | 0 | 1 | 1 | 1 | 0
Extremity necrosis (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Haematoma (Vascular disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypertensive crisis (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Hypovolaemic shock (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Infarction (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Peripheral artery stenosis (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Peripheral embolism (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Peripheral ischaemia (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Shock (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Subclavian vein thrombosis (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Superficial vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Superior vena cava occlusion (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Superior vena cava syndrome (Vascular disorders) | 2 | 2 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Thrombosis (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vasculitis (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Vena cava thrombosis (Vascular disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Venous thrombosis (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Venous thrombosis limb (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1-Arm B: Nivo + Ipi (N=391) | Part 1-Arm A: Nivolumab (N=391) | Part 1-Arm C: Chemotherapy (N=387) | Part 1-Arm D: Nivo + Ipi (N=185) | Part 1-Arm G: Nivo + Chemo (N=172) | Part 1-Arm F: Chemotherapy (N=183) | Part 2 - Arm H: Nivolumab + Chemotherapy (N=375) | Part 2 - Arm I: Chemotherapy (N=371) | Part 3 -Arm J: Nivolumab + Ipilimumab (N=126) | Part 3 - Arm K: Chemotherapy (N=123)
Anaemia (Blood and lymphatic system disorders) | 47 | 51 | 159 | 25 | 80 | 76 | 174 | 151 | 63 | 93
Leukocytosis (Blood and lymphatic system disorders) | 6 | 4 | 1 | 4 | 1 | 1 | 4 | 4 | 9 | 4
Leukopenia (Blood and lymphatic system disorders) | 0 | 3 | 21 | 1 | 10 | 9 | 19 | 15 | 5 | 25
Neutropenia (Blood and lymphatic system disorders) | 4 | 7 | 70 | 2 | 45 | 37 | 66 | 58 | 2 | 16
Thrombocytopenia (Blood and lymphatic system disorders) | 6 | 7 | 39 | 2 | 17 | 14 | 48 | 31 | 2 | 14
Hyperthyroidism (Endocrine disorders) | 33 | 18 | 7 | 19 | 9 | 0 | 11 | 6 | 20 | 3
Hypothyroidism (Endocrine disorders) | 61 | 30 | 4 | 22 | 9 | 1 | 33 | 4 | 27 | 3
Lacrimation increased (Eye disorders) | 3 | 1 | 18 | 1 | 9 | 2 | 20 | 10 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 30 | 30 | 21 | 9 | 10 | 7 | 30 | 15 | 7 | 4
Abdominal pain upper (Gastrointestinal disorders) | 18 | 16 | 22 | 4 | 5 | 6 | 22 | 13 | 8 | 2
Constipation (Gastrointestinal disorders) | 78 | 70 | 104 | 36 | 63 | 53 | 84 | 83 | 20 | 25
Diarrhoea (Gastrointestinal disorders) | 102 | 88 | 66 | 44 | 38 | 33 | 79 | 48 | 26 | 8
Dry mouth (Gastrointestinal disorders) | 17 | 11 | 3 | 6 | 2 | 0 | 11 | 5 | 8 | 0
Dyspepsia (Gastrointestinal disorders) | 15 | 10 | 10 | 7 | 13 | 6 | 12 | 8 | 2 | 0
Mouth ulceration (Gastrointestinal disorders) | 4 | 0 | 3 | 0 | 0 | 0 | 2 | 2 | 8 | 1
Nausea (Gastrointestinal disorders) | 93 | 81 | 174 | 41 | 79 | 74 | 126 | 133 | 17 | 30
Stomatitis (Gastrointestinal disorders) | 25 | 12 | 28 | 2 | 16 | 11 | 17 | 10 | 1 | 3
Vomiting (Gastrointestinal disorders) | 52 | 41 | 73 | 27 | 33 | 34 | 55 | 56 | 20 | 25
Asthenia (General disorders) | 93 | 78 | 66 | 40 | 35 | 42 | 70 | 52 | 17 | 11
Chest discomfort (General disorders) | 4 | 3 | 3 | 2 | 3 | 0 | 6 | 7 | 14 | 7
Chest pain (General disorders) | 19 | 18 | 13 | 4 | 6 | 12 | 16 | 14 | 5 | 3
Fatigue (General disorders) | 107 | 88 | 101 | 38 | 54 | 50 | 87 | 80 | 18 | 23
Malaise (General disorders) | 11 | 13 | 17 | 7 | 13 | 11 | 20 | 24 | 12 | 13
Mucosal inflammation (General disorders) | 13 | 12 | 12 | 3 | 13 | 13 | 19 | 12 | 0 | 0
Non-cardiac chest pain (General disorders) | 16 | 20 | 21 | 17 | 9 | 12 | 18 | 9 | 15 | 12
Oedema peripheral (General disorders) | 49 | 26 | 37 | 18 | 27 | 23 | 40 | 38 | 10 | 4
Pain (General disorders) | 6 | 6 | 6 | 6 | 6 | 4 | 7 | 4 | 10 | 4
Pyrexia (General disorders) | 74 | 57 | 38 | 32 | 33 | 32 | 54 | 38 | 40 | 17
Hepatic function abnormal (Hepatobiliary disorders) | 3 | 0 | 1 | 1 | 2 | 2 | 3 | 2 | 8 | 9
Bronchitis (Infections and infestations) | 17 | 11 | 9 | 9 | 9 | 8 | 18 | 7 | 2 | 0
Nasopharyngitis (Infections and infestations) | 27 | 23 | 22 | 9 | 15 | 4 | 14 | 12 | 1 | 1
Pneumonia (Infections and infestations) | 21 | 20 | 17 | 12 | 10 | 7 | 23 | 27 | 16 | 11
Upper respiratory tract infection (Infections and infestations) | 14 | 17 | 12 | 7 | 14 | 6 | 25 | 14 | 16 | 11
Fall (Injury, poisoning and procedural complications) | 12 | 6 | 2 | 3 | 10 | 1 | 8 | 5 | 0 | 0
Alanine aminotransferase increased (Investigations) | 43 | 40 | 27 | 31 | 22 | 15 | 48 | 29 | 42 | 36
Amylase increased (Investigations) | 30 | 22 | 12 | 18 | 17 | 4 | 33 | 17 | 24 | 4
Aspartate aminotransferase increased (Investigations) | 47 | 37 | 21 | 27 | 16 | 12 | 48 | 25 | 46 | 32
Bilirubin conjugated increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 0 | 14 | 3
Blood alkaline phosphatase increased (Investigations) | 21 | 13 | 12 | 13 | 7 | 4 | 23 | 9 | 18 | 8
Blood bilirubin increased (Investigations) | 5 | 5 | 3 | 3 | 0 | 2 | 9 | 0 | 23 | 10
Blood creatinine increased (Investigations) | 23 | 15 | 21 | 13 | 18 | 10 | 41 | 29 | 13 | 11
Blood glucose increased (Investigations) | 2 | 2 | 3 | 1 | 1 | 0 | 5 | 1 | 7 | 7
Blood lactate dehydrogenase increased (Investigations) | 3 | 5 | 4 | 4 | 2 | 2 | 10 | 5 | 11 | 8
Blood thyroid stimulating hormone decreased (Investigations) | 5 | 3 | 0 | 2 | 1 | 0 | 4 | 0 | 7 | 0
Blood thyroid stimulating hormone increased (Investigations) | 10 | 6 | 3 | 3 | 4 | 1 | 5 | 1 | 7 | 1
Gamma-glutamyltransferase increased (Investigations) | 6 | 7 | 9 | 5 | 2 | 7 | 17 | 10 | 23 | 16
Lipase increased (Investigations) | 31 | 27 | 14 | 25 | 12 | 1 | 27 | 16 | 15 | 6
Lymphocyte count decreased (Investigations) | 7 | 4 | 9 | 2 | 8 | 4 | 3 | 3 | 10 | 9
Neutrophil count decreased (Investigations) | 9 | 11 | 50 | 2 | 31 | 20 | 52 | 54 | 16 | 54
Neutrophil count increased (Investigations) | 1 | 1 | 0 | 0 | 0 | 0 | 4 | 1 | 8 | 3
Platelet count decreased (Investigations) | 6 | 10 | 31 | 2 | 22 | 25 | 38 | 30 | 22 | 49
Weight decreased (Investigations) | 37 | 20 | 22 | 17 | 14 | 8 | 32 | 31 | 44 | 19
Weight increased (Investigations) | 8 | 8 | 3 | 1 | 3 | 1 | 10 | 3 | 7 | 10
White blood cell count decreased (Investigations) | 8 | 5 | 19 | 1 | 17 | 6 | 41 | 39 | 22 | 59
Decreased appetite (Metabolism and nutrition disorders) | 130 | 97 | 109 | 61 | 61 | 52 | 105 | 88 | 40 | 34
Hyperglycaemia (Metabolism and nutrition disorders) | 24 | 16 | 14 | 9 | 6 | 9 | 29 | 20 | 18 | 13
Hyperkalaemia (Metabolism and nutrition disorders) | 10 | 12 | 9 | 6 | 11 | 3 | 12 | 11 | 6 | 5
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 7 | 2
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 8 | 9
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 3 | 1 | 2 | 1 | 2 | 7 | 7 | 20 | 9
Hypoalbuminaemia (Metabolism and nutrition disorders) | 25 | 16 | 14 | 9 | 8 | 7 | 25 | 15 | 41 | 20
Hypocalcaemia (Metabolism and nutrition disorders) | 12 | 9 | 9 | 5 | 7 | 3 | 7 | 6 | 14 | 8
Hypochloraemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 5 | 1 | 17 | 9
Hypokalaemia (Metabolism and nutrition disorders) | 27 | 16 | 12 | 13 | 13 | 9 | 27 | 21 | 24 | 11
Hypomagnesaemia (Metabolism and nutrition disorders) | 12 | 7 | 21 | 10 | 15 | 12 | 25 | 22 | 10 | 6
Hyponatraemia (Metabolism and nutrition disorders) | 39 | 17 | 20 | 14 | 11 | 8 | 25 | 16 | 47 | 18
Hypophosphataemia (Metabolism and nutrition disorders) | 14 | 10 | 11 | 5 | 7 | 5 | 10 | 8 | 8 | 2
Hypoproteinaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 3 | 15 | 14
Arthralgia (Musculoskeletal and connective tissue disorders) | 72 | 62 | 19 | 26 | 28 | 9 | 40 | 40 | 17 | 7
Back pain (Musculoskeletal and connective tissue disorders) | 42 | 36 | 31 | 28 | 23 | 13 | 38 | 29 | 10 | 11
Myalgia (Musculoskeletal and connective tissue disorders) | 23 | 22 | 9 | 9 | 10 | 3 | 30 | 21 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 17 | 24 | 10 | 7 | 14 | 4 | 25 | 21 | 7 | 4
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 9 | 18 | 11 | 5 | 9 | 2 | 12 | 12 | 3 | 2
Dizziness (Nervous system disorders) | 30 | 21 | 27 | 16 | 18 | 21 | 31 | 18 | 16 | 10
Dysgeusia (Nervous system disorders) | 14 | 10 | 25 | 5 | 11 | 9 | 17 | 14 | 0 | 0
Headache (Nervous system disorders) | 54 | 40 | 31 | 13 | 19 | 8 | 34 | 24 | 12 | 8
Neuropathy peripheral (Nervous system disorders) | 1 | 5 | 11 | 2 | 4 | 3 | 26 | 12 | 1 | 0
Paraesthesia (Nervous system disorders) | 14 | 2 | 9 | 4 | 10 | 5 | 19 | 16 | 0 | 0
Anxiety (Psychiatric disorders) | 22 | 12 | 19 | 5 | 7 | 6 | 9 | 13 | 1 | 2
Insomnia (Psychiatric disorders) | 43 | 32 | 30 | 23 | 25 | 11 | 31 | 23 | 22 | 11
Cough (Respiratory, thoracic and mediastinal disorders) | 75 | 82 | 45 | 31 | 45 | 27 | 69 | 44 | 30 | 18
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 98 | 93 | 61 | 47 | 40 | 39 | 74 | 55 | 19 | 16
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 | 9 | 13 | 3 | 9 | 6 | 11 | 9 | 3 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 34 | 26 | 22 | 17 | 9 | 11 | 19 | 20 | 31 | 17
Hiccups (Respiratory, thoracic and mediastinal disorders) | 7 | 10 | 20 | 6 | 9 | 14 | 13 | 13 | 1 | 6
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 22 | 23 | 3 | 6 | 7 | 1 | 16 | 1 | 7 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 28 | 30 | 15 | 12 | 11 | 8 | 24 | 15 | 15 | 14
Alopecia (Skin and subcutaneous tissue disorders) | 8 | 9 | 34 | 3 | 12 | 10 | 45 | 45 | 3 | 5
Dry skin (Skin and subcutaneous tissue disorders) | 37 | 14 | 12 | 9 | 11 | 4 | 7 | 9 | 1 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 92 | 44 | 17 | 29 | 23 | 5 | 38 | 11 | 27 | 5
Rash (Skin and subcutaneous tissue disorders) | 93 | 55 | 31 | 31 | 29 | 13 | 59 | 32 | 32 | 15
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 28 | 13 | 7 | 14 | 9 | 4 | 10 | 4 | 5 | 2
Hypertension (Vascular disorders) | 21 | 15 | 13 | 8 | 12 | 8 | 21 | 8 | 8 | 3
Hypotension (Vascular disorders) | 16 | 13 | 9 | 6 | 10 | 8 | 9 | 8 | 5 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-15): https://cdn.clinicaltrials.gov/large-docs/26/NCT02477826/Prot_SAP_000.pdf